CLINICAL TRIAL: NCT00873808
Title: Long-Term Bone Quality in Women With Breast Cancer (A Companion Study to S0307)
Brief Title: S0307A, Long-Term Bone Quality in Women With Breast Cancer Enrolled on Clinical Trial SWOG-S0307
Status: Withdrawn | Type: Observational
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000614118; S0307A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Clodronic Acid; Demeclocycline; Ibandronic Acid; Tetracycline; Zoledronic Acid; Chemotherapy, Adjuvant; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: clodronate disodium
Drug: demeclocycline hydrochloride
Drug: ibandronate sodium
Drug: tetracycline hydrochloride
Drug: zoledronic acid
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: computed tomography
Procedure: dual x-ray absorptiometry

SUMMARY:
RATIONALE: Gathering information over time from imaging and laboratory tests of women receiving bisphosphonates for breast cancer may help doctors learn more about long-term bone quality and plan the best treatment. Tetracycline hydrochloride and demeclocycline hydrochloride can mark the new growth of the bone, so it may be seen better under a microscope.

PURPOSE: This clinical trial is studying long-term bone quality in women with breast cancer enrolled on clinical trial SWOG-S0307.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess if long-term high-dose bisphosphonates alter bone quality as measured by change in the histomorphometry of bone biopsies after tetracycline hydrochloride labeling to calculate eroded and osteoid surfaces, mineralization surface, bone formation rate, wall width, and activation frequency.
* To assess if long-term high-dose bisphosphonates alter bone quality as measured by change in the backscattered electron imaging of bone to measure average mineralization density as well as distribution of density values.
* To assess if long-term high-dose bisphosphonates alter bone quality as measured by change in the micro-computed tomography of bone biopsy specimens to measure bone structure, including bone volume, connectivity, trabecular width, and cortical width.
* To assess if long-term high-dose bisphosphonates alter bone quality as measured by change in the biomechanical testing of bone biopsy samples loaded in compression to measure stress-strain relationships, including Young's modulus, yield point, ultimate strain, and work to failure (toughness).
* To characterize bone using classical, non-invasive techniques (i.e., measurement of bone mineral density of spine and hip using dual energy x-ray absorptiometry and analysis of serum biochemical markers of bone formation [i.e., bone specific alkaline phosphatase] and resorption [i.e., N-telopeptide]) after long-term, high-dose bisphosphonates.

OUTLINE: This is a multicenter study.

At baseline (prior to initiating bisphosphonate therapy on SWOG-S0307), patients receive oral tetracycline hydrochloride twice daily on days 1 and 2 and oral demeclocycline hydrochloride twice daily on days 11 and 12. Patients undergo a tetracycline hydrochloride-labeled bone biopsy from the anterior ilium on day 14. At 36 months (for patients who have completed bisphosphonate therapy) or after 30 months of concurrent bisphosphonate therapy, patients receive oral demeclocycline twice daily on days 1 and 2 and oral tetracycline hydrochloride twice daily on days 11 and 12. Patients undergo a demeclocycline hydrochloride-labeled bone biopsy from the anterior ilium on day 14.

Patients undergo dual energy x-ray absorptiometry measurements of the hip and spine at the time of biopsy or within the next 10 weeks. Blood samples are collected for analysis of bone specific alkaline phosphatase and N-telopeptide before and after treatment on the clinical trial.

After completion of study treatment, patients are followed for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Concurrently enrolled on clinical trial SWOG-S0307 and receiving bisphosphonates as adjuvant therapy for primary breast cancer
* No rickets, osteogenesis imperfecta, osteosclerosis, or osteomalacia
* No bone fracture since the age of 21 years unless it was caused by trauma
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Weight < 300 lbs
* No hyperparathyroidism
* No serious concurrent or prior anorexia nervosa diagnosed by a physician and causing abnormal menstruation
* No history of hypersensitivity to tetracycline or demeclocycline

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 10 years since prior prednisone at a dose above 5 mg/day for ≥ 3 months
* No prior prednisone before diagnosis of breast cancer
* No prior bisphosphonate therapy
* No concurrent anticonvulsant medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in bone quality after long-term high-dose bisphosphonates as measured by histomorphometry, mineralization density, micro-computed tomography, and biomechanics of bone biopsy samples

SECONDARY OUTCOMES:
Comparison of the potency of bisphosphonates as measured by changes in bone quality in each treatment group
Correlations among measures of bone formation, structure, mineralization, and strength

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- University Cancer Center at University of Washington Medical Center, Seattle, Washington, United States